CLINICAL TRIAL: NCT06252987
Title: The Second Hospital of Dalian Medical University
Brief Title: The Effects of tDCS Combined With rTMS on Post-stroke Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fnirs
Record Dates: First submitted 2024-01-17; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- common group (Sham Comparator): routine training
  Interventions: Other: routine treatment
- tDCS group (Experimental): tDCS
  Interventions: Other: routine treatment; Other: Non-invasive brain stimulation
- rTMS group (Experimental): rTMS
  Interventions: Other: routine treatment; Other: Non-invasive brain stimulation
- Combination group (Experimental): tDCS-rTMS
  Interventions: Other: routine treatment; Other: Non-invasive brain stimulation

INTERVENTIONS:
Other: routine treatment — Routine medical treatment, basic rehabilitation training and individualized cognitive training
Other: Non-invasive brain stimulation — tDCS&rTMS
  Arms: Combination group; rTMS group; tDCS group

SUMMARY:
If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects]

The purpose of the clinical trial is to find a treatment for stroke patients with cognitive impairment, and the main questions it aims to answer are:

* [Search for effective treatments of cognitive impairment after stroke]
* [Explore brain network features with functional near-infrared spectroscopy] Participants will receive conventional treatment, tDCS treatment, or rTMS treatment, or tDCS-rTMS treatment.

And then compare cognitive function and brain function.

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical diagnostic criteria of the Expert Consensus on the Management of Cognitive Impairment after Stroke in 2021;
* 30-80 years old, right-handed, unilateral hemiplegia;
* Verbal expression can cooperate with the completion of the evaluation, sustained attention time is longer than 5 minutes;
* Simple Mental State Examination Scale (MMSE) score ≤26 points; MoCA scale score < 26 points; Memory test (RMBT) score less than 21 points;
* patients or their family agree to sign the informed consent;
* The Ethics Committee approved the trial.

Exclusion Criteria:

* Memory dysfunction caused by other diseases, such as Alzheimer's disease, lewy body dementia, pituitary tumor surgery, hypothyroidism, etc.;
* There are contraindications of rTMS and tDCS for untreated intracranial aneurysms, severe epilepsy, intracranial metal, etc.
* Patients with severe visual, cognitive or speech impairment who cannot cooperate with treatment;
* The condition is not stable; Or other serious physical diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of brain's HbO by functional near-infrared spectroscopy | 2 weeks
  fNIRS

SECONDARY OUTCOMES:
Score of Mini-Mental State Examination | 2 weeks
  MMSE
Score of The Frontal Assessment Battery | 2 weeks
  FAB
Score of Attention assessment by the digit span task | 2 weeks
  DST

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Jiang, Study Director — Department of Rehabilitation Medicine, the Second Hospital of Dalian Medical University
Locations (1):
- Lily, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No